CLINICAL TRIAL: NCT02105779
Title: Optimizing Cognitive Remediation Outcomes in Schizophrenia
Acronym: CAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01MH082818 (NIH)
Record Dates: First submitted 2014-03-11; First posted 2014-04-07 (Estimated); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Schizophrenia; Psychosis
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Targeted Cognitive Training (Experimental): 40 hours of BFP auditory training
  Interventions: Other: Targeted Cognitive Training
- Social Cognitive Training (Experimental): 40 hours of auditory training and 10 hours social exercises
  Interventions: Other: Social Cognitive Training

INTERVENTIONS:
Other: Targeted Cognitive Training — At present, the TCT exercises consist of three modules: an Auditory Processing Module (40-50 hours of training); a Visual Processing Module (30 hours); a Cognitive Control Module prototype (20 hours). [Based on the results of our current RCT, Posit Science has revised aspects of the training modules in order to further optimize its effectiveness for treatment of schizophrenia. In this study, we will use updated versions of the training software: an Auditory Module (30 hours), and a Visual Module (30 hours). Features from the Cognitive Control module prototype have been expanded and incorporated into these new modules.
  Arms: Targeted Cognitive Training
Other: Social Cognitive Training — We developed a systematic approach to basic training in facial emotion identification and discrimination and simple social perception and theory of mind tasks using components drawn from three commercially available software packages: the MicroExpressions Training Tool and The Subtle Expressions Training Tool (METT and SETT), plus the MindReading program. Training begins with simple emotion identification tasks, and slowly progressed to more difficult tasks that required subjects to discriminate between two subtle emotion expressions, and to correctly interpret the emotional significance of brief social scenes. A total of 10 hours of training occurred over 8 weeks.
  Arms: Social Cognitive Training

SUMMARY:
The purpose of this study is to drive an optimal response to neuroplasticity-based cognitive remediation in schizophrenia in order to maximize treatment response. The investigators will investigate factors that have generally been ignored in prior computer-based cognitive remediation programs-those related to social cognition-- and will delineate their relationship to motivation, functional outcome, and the neural substrates of reward anticipation and emotion processing. Current research indicates that, unless the investigators fully understand and harness these factors, the investigators will not achieve meaningful treatment gains for individuals with schizophrenia.

DETAILED DESCRIPTION:
The purpose of this study is to explicitly and aggressively drive an optimal response to neuroplasticity- based cognitive remediation in schizophrenia in order to maximize treatment response. We will investigate factors that have generally been ignored in computer-based cognitive remediation programs-those related to social cognition-- and will delineate their relationship to motivation, functional outcome, and the neural substrates of reward anticipation and emotion processing. Current research indicates that, unless we fully understand and harness these factors, we will not achieve meaningful treatment gains for individuals with schizophrenia.

Our specific aims are:

1. To perform an RCT in which 100 schizophrenia subjects are assigned to either 60 hours of neuroplasticity- based computerized targeted cognitive training (TCT) that focuses exclusively on "cold cognition" (a program which trains early sensory processing, attention, working memory and cognitive control in auditory and visual domains), or to 60 hours of training that combines the TCT program with 20 minutes per day of adaptive computerized social cognition training (SCT) exercises.
2. To compare the outcomes of these two groups of subjects on measures of neurocognition, social cognition, motivation, and functional outcome.
3. To assess subjects six months after the intervention to determine the durability of training effects.
4. To identify changes in brain activation patterns in key neural regions as a result of TCT alone vs. TCT+SCT: during reward anticipation, and during emotion recognition.

The timeliness of this approach is supported by recent evidence demonstrating only weak associations between traditional cognitive remediation approaches and functional outcome in schizophrenia, but a strong, direct relationship between social cognition and functional outcome. Thus we must now examine the clinical, functional, and neural effects of a well-designed state-of-the-art cognitive training program that combines neurocognition with social cognition training.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of schizophrenia or schizoaffective disorder
* Between 18-65 years of age
* Clinically stable
* Fluent in English

Exclusion Criteria:

* Recent hospitalization, in the past 3 months
* History of traumatic brain injury
* Neurological disorders
* Inability to participate in the study soberly

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2009-12; Primary Completion 2016-05 (Actual); Study Completion 2016-07-26 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Social Cognition at 6 months | Baseline (Intake)/6 months follow-up after trianing completion
  Social functioning scale

CONTACTS AND LOCATIONS:
Overall Officials: Sophia Vinogradov, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco Veterans Medical Center, San Francisco, California, United States

REFERENCES:
- [Derived] Fisher M, Nahum M, Howard E, Rowlands A, Brandrett B, Kermott A, Woolley J, Vinogradov S. Supplementing intensive targeted computerized cognitive training with social cognitive exercises for people with schizophrenia: An interim report. Psychiatr Rehabil J. 2017 Mar;40(1):21-32. doi: 10.1037/prj0000244. PMID 28368179
- [Derived] Biagianti B, Fisher M, Neilands TB, Loewy R, Vinogradov S. Engagement with the auditory processing system during targeted auditory cognitive training mediates changes in cognitive outcomes in individuals with schizophrenia. Neuropsychology. 2016 Nov;30(8):998-1008. doi: 10.1037/neu0000311. Epub 2016 Sep 12. PMID 27617637